CLINICAL TRIAL: NCT04935697
Title: Non-invasive Vagal Neurostimulation (nVNS) to Mitigate Traumatic Brain Injury (TBI)-Induced Acute Respiratory Distress and Acute Lung Injury
Brief Title: Non-invasive Vagal Neurostimulation (nVNS) for Traumatic Brain Injury (TBI)-Induced Acute Respiratory Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: ElectroCore INC (Industry); Chuck Noll Foundation (Unknown)
Responsible Party: Principal Investigator, Edward Snell, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nVNS for TBI-ALI/ARDS
Record Dates: First submitted 2021-03-12; First posted 2021-06-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury; Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS); Traumatic Brain Injury
Keywords: Non-invasive Vagal Nerve Stimulation
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Receiving Non-invasive vagus neurostimulation (Experimental): nVNS treatment will be applied three times daily. One treatment is defined as 2 consecutive stimulations: one, 2-minute stimulation on the side of the neck followed by a second, 2-minute stimulation on the same side of the neck. The treatment will be done 3 times per day (morning, mid-day and 1 hour before bed at night), every day, until patient is discharged from the hospital or requires mechanical ventilation. Patient will record the time they administered these treatments. If the patient is unable to do this, a research staff member who has been trained on the device can assist. Will also receive SOC for TBI.
  Interventions: Device: nVNS; Other: SOC
- Receiving Standard of Care (Other): Patients will be managed according to the institutional best practices and SOC for TBI.
  Interventions: Other: SOC

INTERVENTIONS:
Device: nVNS — 3x daily treatment of nVNS + SOC
  Arms: Receiving Non-invasive vagus neurostimulation
Other: SOC — Standard of care patient management.

SUMMARY:
This is a prospective, randomized, two-arm, controlled 30-day investigational pilot trial using the gammaCore Sapphire S non-invasive vagus nerve stimulation (nVNS) device + standard of care (SOC) in newly-hospitalized patients with mild-to-moderate traumatic brain injury (TBI) to prevent the progression towards immunokine storms, systemic inflammatory response syndrome (SIRS), severe respiratory distress, and requirement for invasive mechanical ventilation, and death, when compared to SOC alone (the control arm).

DETAILED DESCRIPTION:
A pilot population of 46 individuals between 18-80 years of age inclusive, will be enrolled, with an in-trial monitoring period of up to 30 days following baseline measurements. Study subjects will remain in-trial until one of the following occurs: a) 30 days without any progression to respiratory distress requiring mechanical ventilation; b) requirement for mechanical ventilation prior to 30 days; or c) death prior to 30 days. In addition to the screening, a total of up to 5 additional in-trial events (depending on the time at discharge from hospitalization) plus one additional clinical site visit at the end of the follow-up period will comprise the study events schedule of this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 12-80 years, inclusive
2. Patient has been admitted to the hospital for mild-to-moderate TBI that is restricted to the head and/or neck region.
3. Patient is not on invasive mechanical ventilation
4. Patient has a mild-to-moderate TBI based on a non-resuscitated or post-resuscitated Glasgow Coma Scale (GCS) sum score of =>12
5. Patient has a Lung Injury Prediction Score (LIPS) of =>2
6. Administration of the first nVNS treatment must be planned to take place within 24 h of intake
7. A signed, written informed consent form from the patient or legally authorized representative

Exclusion Criteria:

1. Patient has a diagnosis of moderate or greater grade of respiratory distress/ARDS according to the Berlin definition of ARDS: Partial pressure of oxygen (PaO2) /Fraction of Inspired Oxygen (FiO2) > 100 mmHg (>13.3 kPa) to ≤ 200 mmHg (≤ 26.6 kPa) with positive end-expiratory pressure (PEEP) ≥ 5 cmH2O)
2. Woman known to be pregnant, lactating or with a positive (urine or serum test) or indeterminate (serum test) pregnancy test
3. Patient simultaneously taking part in another clinical trial
4. Patient is not expected to survive for 24 hours
5. Patient has an underlying clinical condition where, in the opinion of the study physicians and the institutional health provider physician, it would be extremely unlikely that the patient would not progress to invasive mechanical ventilation within 48 hours or any other condition that might require immediate invasive mechanical ventilation (e.g. motor neuron disease, Duchenne muscular dystrophy, or rapidly-progressive interstitial pulmonary fibrosis)
6. Patient has severe chronic obstructive pulmonary disease (COPD) requiring long-term home oxygen therapy or mechanical ventilation (non-invasive ventilation or via tracheotomy) except for continuous positive airway pressure (CPAP) or bi-level positive airway pressure (BIPAP) used solely for sleep-disorder breathing
7. Patient has congestive heart failure
8. Patient has acute left ventricular failure
9. Patient has liver failure (Child-Pugh grade C)
10. Patient is receiving renal dialysis therapy for chronic renal failure
11. Patient is receiving extracorporeal membrane oxygenation, high-frequency oscillatory ventilation (HFOV) or any form of extracorporeal lung support
12. Patient has had any form of mechanical ventilation (invasive or non-invasive, excluding CPAP alone) for longer than 48 h prior to the diagnosis of mild-to-moderate respiratory distress/ARDS
13. Patient has burns to ≥ 15% of their total body surface area

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Days free of invasive mechanical ventilation | 30 days from baseline
  Days free of invasive mechanical ventilation within 30 days from baseline among TBI survivors.
Days free of death | 30 days from baseline
  Days free of death within 30 days from baseline

SECONDARY OUTCOMES:
Adverse Events/Serious Adverse Events (AEs/SAEs) | Day 30 from baseline, Day 60, Day 90
  Incidence, rate and severity of AEs/SAEs
Incidence of abnormal Physical examinations | Day 30 from baseline or last day in hospital, Day 60, Day 90
  Physical examination results
Incidence of abnormal vital signs | Day 30 from baseline or last day in hospital, Day 60, Day 90
  vital sign results
Incidence of abnormal laboratory results | Day 30 from baseline or last day in hospital, Day 60, Day 90
  laboratory results
All-cause mortality | Day 30 from baseline, Day 60, Day 90
  All-cause mortality
Days free of organ failure | Day 30 from baseline or last day in study, Day 60, Day 90
  assessed using the Sequential Organ Failure Assessment (SOFA) score (numerically quantifies (0-4) the number and severity of failed organs) with higher number being worse
Days free of renal support | Day 30 from baseline or last day in study
Days free of vasoactive support | Day 30 from baseline or last day in study
Number of ICU-free days | Day 30 from baseline
  assessed at Day 30 or on the last day in the ICU if the patient leaves the ICU before Day 30
Days free of invasive mechanical ventilation | Day 30 from baseline of last day in study
Length of hospital stay | Study Completion (up to 95 days from baseline)
  Number of days in hospital
Forced Expiratory Volume (FEV1) | Day 30 from baseline, Day 60 from baseline, Day 90 from baseline
Neurological functioning | Day 30 from baseline, Day 60 from baseline, Day 90 from baseline
  6 minute walk test
PROMIS CAT score (Patient-Reported Outcomes Measurement Information System (PROMIS) computer adaptive testing (CAT)) | Day 30 from baseline, Day 60 from baseline, Day 90 from baseline
  0 to 100, with 0 being the lowest physical function and most disabled and 100 having the highest functioning
Post concussion symptom scale (PCSS) | Day 30 from baseline, Day 60 from baseline, Day 90 from baseline
  27 perceived symptoms, patient reports their current experience of symptoms, on a scale from 0 to 6, with 0 being "none/not experiencing particular symptom" to 6 being experiencing "severe" symptom; total point value of scale is from 0 to 162

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kimutis, Study Director — Allegheny Health Network
Locations (1):
- AHN Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No